CLINICAL TRIAL: NCT01426191
Title: A Open Multi-center Clinical Study on Cefotaxime Sodium and Sulbactam Sodium for Injection(2:1) for Treatment of Respiratory and Urinary Tract Infection
Brief Title: Study on Cefotaxime and Sulbactam Sodium for Injection (2:1) for Treatment of Respiratory and Urinary Tract Infection
Acronym: SWSB
Status: Completed | Type: Observational
Sponsor: Xiangbei Welman Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 20090095
Record Dates: First submitted 2011-08-23; First posted 2011-08-31 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Respiratory Tract Infections; Urinary Tract Infections
Keywords: Cefotaxime sulbactam sodium; Phase IV clinical studies; Respiratory and urinary tract infections
MeSH Terms: conditions — Respiratory Tract Infections; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- xinzhijun: 1.5-3.0g,iv,bid or tid for 5-12 days
  Interventions: Drug: xinzhijun

INTERVENTIONS:
Drug: xinzhijun — durg:Cefotaxime sodium and sulbactam sodium for injection(2:1)
  1.5-3.0g,iv,bid or tid for 5-12 days;
  Serious infections:1.0-1.5g,iv,tid or qid for 5-12 days
  Other Names: Experimental; shumate

SUMMARY:
In the proposed study, the investigators plan to evaluate the efficacy and safety of Cefotaxime sodium and sulbactam sodium for injection (2:1)for the treatment of respiratory and urinary tract acute bacterial infection under the widely used in clinical conditions.

DETAILED DESCRIPTION:
Cefotaxime is a third-generation cephalosporins.Cefotaxime sodium and sulbactam sodium for injection (2:1)plays a therapeutic role by the former inhibiting bacterial cell wall synthesis by irreversible competitive inhibition of β-lactamase.The antimicrobial effect of cefotaxime can be enhanced by the two combined.The compound specifically aims to the mechanism of bacterial resistance, extending the life of cefotaxime in the treatment-resistant pathogen infections.

ELIGIBILITY:
Inclusion Criteria:

1. patients who qualify for moderate and severe acute respiratory or urinary tract bacterial infection of acute bacterial infections need for systemic antibiotic therapy.
2. Age>18 years old, Gender: both
3. Women of childbearing age were to be negative pregnancy test and agree to take contraceptive measures during the trial;
4. patients were volunteers and signed informed consent form;
5. patients did not participate in other clinical trials.

Exclusion Criteria:

1. Patients were hypersusceptibility to the test drug or other penicillins ,β-lactamase inhibitor
2. Pregnant and Lactating women
3. Patients have severe liver,kidney,cardiovascular,cerebrovascular,endocrine and hematopoietic system of primary diseases and that of immunodeficiency,advanced cancer or mental illness.
4. Patients who were complicated by other diseases and thought to affect efficacy evaluations or poor compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalized patients or outpatients
Sampling Method: Non-Probability Sample
Enrollment: 2032 (Actual)
Dates: Start 2011-08; Primary Completion 2015-04 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: lanjuan lj li, docter, Principal Investigator — Zhejiang University; changqing cq li, doctor, Study Director — Chongqing Red Cross Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: post market
Pre-assignment Details: Third-generation cephalosporin resistant
Groups:
- Xinzhijun: 1.5-3.0g,iv,bid or tid for 5-12 days
  xinzhijun: durg:Cefotaxime sodium and sulbactam sodium for injection(2:1)
  1.5-3.0g,iv,bid or tid for 5-12 days;
  Serious infections:1.0-1.5g,iv,tid or qid for 5-12 days
Period: Overall Study
Arm/Group | Xinzhijun
Started | 2032
Completed | 2032
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Xinzhijun: xinzhijun:third generation beta-lactam cephalosporin and beta lactamase inhibitors (BLIs)
Arm/Group | Xinzhijun
Number analyzed (Participants) | 2032
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1982
  >=65 years | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1250
  Male | 782
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Chinese: American Indian or Alaska Native | 0
  Chinese: Asian | 2032
  Chinese: Native Hawaiian or Other Pacific Islander | 0
  Chinese: Black or African American | 0
  Chinese: White | 0
  Chinese: More than one race | 0
  Chinese: Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 2032

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: the incidence(%)of allergies, skin rashes, shock,death, etc.
Time Frame: day0-day22-28
Measure: Count of Participants; unit: Participants
Arm/Group | Xinzhijun
Number analyzed (Participants) | 2032
Participants
  nausea | 10
  vomiting | 4
  diarrhea | 6
  Pyrexia | 10
  ALT increased | 25
  AST increased | 15
  no | 1962
Statistical Analysis 1: Comparison: Xinzhijun; Test type: Other; p = 0.05, Fisher Exact

2. Secondary Outcome: Clinical Effect
Description: outcome:1.clinical cure 2. clinical failure population included patients who received the study drug, complied with the study protocol, did not have a missing or indeterminate clinical outcome response at the test-of-cure (TOC) visit, and had no confounding factors that interfered with the assessment of clinical outcome (e.g., use of nonstudy systemic antibiotic therapy on or after the first dose of the study drug for reasons other than treatment failure).
Time Frame: at weeks 4,day22-28
Population: included all the participants
Measure: Count of Participants; unit: Participants
Arm/Group | Xinzhijun
Number analyzed (Participants) | 2032
Participants
  cure | 2022
  failure | 10
Statistical Analysis 1: Comparison: Xinzhijun; Test type: Other; p = 0.01, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Xinzhijun
All-Cause Mortality (participants affected / at risk) | 0/2032
Serious Adverse Events (participants affected / at risk) | 0/2032
Other Adverse Events (participants affected / at risk) | 70/2032
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xinzhijun (N=2032)
nausea (Gastrointestinal disorders) | 10 (10)
vomiting (Gastrointestinal disorders) | 4 (4)
diarrhea (Gastrointestinal disorders) | 6 (7)
pyrexia (Nervous system disorders) | 10 (11)
ALT increased (Blood and lymphatic system disorders) | 25 (25)
AST increaesd (Blood and lymphatic system disorders) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days